CLINICAL TRIAL: NCT00715585
Title: Addressing The Role of Nutrition Education & Health Literacy in Diabetes Care
Acronym: DiNES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: American Association of Diabetes Educators (Other)
Responsible Party: Principal Investigator, Russell Rothman, Prinicipal Investigator, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08335
Record Dates: First submitted 2008-07-10; First posted 2008-07-15 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Diabetes
Keywords: diabetes; education; health literacy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Active Control (Active Comparator): patients receive 3 individualized visits with a health educator for education on general diabetes and health promotion
  Interventions: Behavioral: Active Control
- Intervention 1 (Experimental): patients receive 3 individualized visits with an rd-cde for education focused on modified plate method
  Interventions: Behavioral: int arm 1
- intervention 2 (Experimental): patients receive 3 individualized visits with an rd-cde for education focused on carb counting
  Interventions: Behavioral: int arm 3

INTERVENTIONS:
Behavioral: Active Control — patients receive 3 individualized visits with a health educator focused on general diabetes education and health promotion
  Arms: Active Control
Behavioral: int arm 1 — VVpatients receive 3 individualized visits with an rd-cde for education focused on modified plate method
  Arms: Intervention 1
Behavioral: int arm 3 — patients receive 3 individualized visits with an rd-cde for education focused on carb counting
  Arms: intervention 2

SUMMARY:
This study examines the impact of certified diabetes education, and the role of different educational approaches to medical nutrition therapy. in addition the role of patient health literacy level is assessed

DETAILED DESCRIPTION:
150 patients with type 2 diabetes with most recent a1c>7% will be enrolled. patients are randomized to three arms: arm 1 includes 3 individualized visits with an rd-cde focused on a modified plate method for nutrition therapy, arm 2 includes 3 individualized visits with an rd-cde focused on carb counting for nutrition therapy, and arm 3 focuses on general diabetes education and health promotion. education sessions will be administered over a 4-6 week period. patients will be assessed at baseline, 3 and 6 month follow-up. primary outcome is a1c.

ELIGIBILITY:
Inclusion Criteria:

* Most recent a1c >7
* Type 2 diabetes
* Receiving primary care
* Not currently in the diabetes improvement program
* No plans to refer to diabetes improvement program in the next 6 mos

Exclusion Criteria:

* Significant dementia or psychosis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2008-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
A1C | 6 months

SECONDARY OUTCOMES:
self-efficacy | 3 and 6 months
satisfaction | 3 and 6 months
dietary behavior | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Russell Rothman, MD MPP, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt, Nashville, Tennessee, United States